CLINICAL TRIAL: NCT00486863
Title: S. Japonicum and Pregnancy Outcomes: A Randomized, Double Blind, Placebo Controlled Trial (RCT)
Brief Title: S. Japonicum and Pregnancy Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-0039
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2014-07

CONDITIONS: Schistosomiasis
Keywords: Philippines, Schistosoma japonicum, Schistosomiasis, pregnant women, fetuses, 08-0049
MeSH Terms: conditions — Schistosomiasis; Schistosomiasis japonica | interventions — Praziquantel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Control (Placebo Comparator): Placebo at 12-16 weeks gestation.
  Interventions: Other: Placebo
- Praziquantel (Experimental): Praziquantel at 12-16 weeks gestation.
  Interventions: Drug: Praziquantel

INTERVENTIONS:
Drug: Praziquantel — 60 mg/kg administered orally given in split dose (30/mg/kg each) separated by 3 hours; over-encapsulated in gelatin capsules. Two capsule sizes will be made which will be differentiated by color; these will contain 300 mg or 150 mg to allow for best dosing by weight.
  Arms: Praziquantel
Other: Placebo — Made with the same color coded gelatin capsules with the inert compound dextrose.
  Arms: Control

SUMMARY:
The purpose of the study is to understand whether the drug praziquantel (PZQ) is safe for the mother and developing baby when the mother has schistosomiasis (a type of worm) infection, and whether the drug may improve the mother's and baby's health. The usual practice is to wait until after a mother has finished breast feeding before giving the medicine. Approximately 375 infected pregnant women, ages 18 and over, in endemic villages in Leyte, The Philippines will participate. Study volunteers 12-16 weeks pregnant will be given PZQ or an inactive pill (placebo) and stay in the hospital overnight. Small blood samples will be collected before and after the medication is taken. Three stool and urine samples will be taken during a total of 7 study visits. An ultrasound image (picture or outline of the unborn baby) will be performed. When the baby is born, a small blood sample will be taken. Mother and baby will be followed for up to 8 months before the baby is born and 1 month after.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled study will investigate praziquantel (PZQ) for the treatment of Schistosomiasis japonicum in pregnant women living in endemic villages of Leyte, The Philippines. The study will enroll 375 pregnant women, ages 18 and over, infected with S. japonicum. The primary study objective is to quantify the efficacy of PZQ treatment for S. japonicum at 12-16 weeks gestation on newborn birth weight among live births. This will be assessed by measuring birth weight within 96 hours of delivery to 10 grams. The secondary objectives are to: 1) assess treatment efficacy with respect to maternal and newborn nutritional status and maternal parasitologic response to treatment; 2) collect preliminary safety and toxicity data on use of PZQ among pregnant women and their newborns; 3) identify extra-placental mechanisms mediating the hypothesized beneficial effect of PZQ on birth outcomes; and 4) identify extra-placental mechanisms mediating the hypothesized beneficial effect of PZQ on birth outcomes. Participants will be involved in study related procedures for 9 months (8 months pre-natally and 1 month post-natally) for mother and infant. This study is linked to DMID protocol 08-0049.

ELIGIBILITY:
Inclusion Criteria:

For screening:

* Female, age 18 or over.
* Present to a study midwife with suspected pregnancy.
* Live in a study village.

For the main study:

* Infected with S. japonicum.
* Pregnancy as determined by urine pregnancy test.
* Age 18 or older.
* Participant is otherwise healthy as determined by history, physical exam, ultrasound and laboratory assessment.
* Pregnancy between 12-16 weeks gestation.
* Ability to provide informed consent to participate.

Exclusion Criteria:

* Presence of significant disease/illness that is either acute or chronic. This will be defined by history, physical examination, ultrasound and laboratory assessment. In particular:

  1. History of seizures or other neurologic disorder, chronic medical problem determined by history or physical examination, e.g. active hepatitis, tuberculosis, heart disease.
  2. Grade 3 or higher laboratory abnormality of blood urea nitrogen (BUN), Creatinine, bilirubin, white blood cell count, or platelet count will warrant exclusion. Grade 2 or higher abnormality of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) will warrant exclusion. For hemoglobin, women with severe anemia defined as hemoglobin less than 7.0 g/dl will be excluded.
  3. Women with myoma on ultrasound that are sub-mucosal or women with myoma that is in any location and greater than 5 cm in size.
  4. Women with congenital anomalies of the reproductive tract that would be expected to cause decreased fetal weight or greatly increase the risk of prematurity such as duplicate uterus, uterine septum.
  5. For less clear cases, the researchers will define significant illness as one that significantly alters a woman's ability to perform activities of daily living, causes symptoms at least two days per week, or necessitates regular use of medication. In the case of acute medical conditions such as urinary tract infection, pneumonia, febrile illness, enrollment may be postponed until the illness is successfully treated (not currently on any medication for the illness) or the illness self resolves if this occurs before 16 weeks gestation.
* Presence of cysts in the eye suggestive of neurocysticercosis.
* Regular use of a medication for a chronic medical condition.
* History of severe allergic reaction (anaphylaxis, facial swelling, or difficulty breathing) or seizure with praziquantel administration.
* Fetus has congenital anomaly determined by 12-16 week ultrasound or is determined to be nonviable (e.g. blighted ovum).
* Twin or higher order pregnancy.
* Woman has been enrolled into this study for a previous pregnancy.
* Inability to comprehend study procedures and provide informed consent due to limited cognitive abilities or other, or refuses to provide informed consent.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2007-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Tropical Medicine - Health Compound, Muntinlupa City, National Capital Region, Philippines

REFERENCES:
- [Derived] Salam RA, Das JK, Bhutta ZA. Effect of mass deworming with antihelminthics for soil-transmitted helminths during pregnancy. Cochrane Database Syst Rev. 2021 May 17;5(5):CD005547. doi: 10.1002/14651858.CD005547.pub4. PMID 33998661
- [Derived] Colt S, Jarilla B, Baltazar P, Tallo V, Acosta LP, Wu HW, Barry CV, Kurtis JD, Olveda RM, Friedman JF, Jiz MA. Effect of maternal praziquantel treatment for Schistosoma japonicum infection on the offspring susceptibility and immunologic response to infection at age six, a cohort study. PLoS Negl Trop Dis. 2021 Apr 16;15(4):e0009328. doi: 10.1371/journal.pntd.0009328. eCollection 2021 Apr. PMID 33861768
- [Derived] Abioye AI, McDonald EA, Park S, Joshi A, Kurtis JD, Wu H, Pond-Tor S, Sharma S, Ernerudh J, Baltazar P, Acosta LP, Olveda RM, Tallo V, Friedman JF. Maternal, placental and cord blood cytokines and the risk of adverse birth outcomes among pregnant women infected with Schistosoma japonicum in the Philippines. PLoS Negl Trop Dis. 2019 Jun 12;13(6):e0007371. doi: 10.1371/journal.pntd.0007371. eCollection 2019 Jun. PMID 31188820
- [Derived] Abioye AI, Park S, Ripp K, McDonald EA, Kurtis JD, Wu H, Pond-Tor S, Sharma S, Ernerudh J, Baltazar P, Acosta LP, Olveda RM, Tallo V, Friedman JF. Anemia of Inflammation during Human Pregnancy Does Not Affect Newborn Iron Endowment. J Nutr. 2018 Mar 1;148(3):427-436. doi: 10.1093/jn/nxx052. PMID 29546300
- [Derived] Blake RA, Park S, Baltazar P, Ayaso EB, Monterde DB, Acosta LP, Olveda RM, Tallo V, Friedman JF. LBW and SGA Impact Longitudinal Growth and Nutritional Status of Filipino Infants. PLoS One. 2016 Jul 21;11(7):e0159461. doi: 10.1371/journal.pone.0159461. eCollection 2016. PMID 27441564
- [Derived] Olveda RM, Acosta LP, Tallo V, Baltazar PI, Lesiguez JL, Estanislao GG, Ayaso EB, Monterde DB, Ida A, Watson N, McDonald EA, Wu HW, Kurtis JD, Friedman JF. Efficacy and safety of praziquantel for the treatment of human schistosomiasis during pregnancy: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2016 Feb;16(2):199-208. doi: 10.1016/S1473-3099(15)00345-X. Epub 2015 Nov 2. PMID 26511959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were otherwise healthy schistosomiasis-infected women at 12-16 weeks gestation, recruited from approximately 50 schistosomiasis-endemic villages served by 6 municipal health centers in Leyte, The Phillipines. Participants were enrolled between 13Aug2007 and 5Nov2012.
Groups:
- Placebo Control at 12-16 Weeks Gestation: Placebo was made with the same color-coded gelatin capsules as the test agent, but with the inert compound dextrose.
- Praziquantel at 12-16 Weeks Gestation: Praziquantel was administered orally as 60 mg/kg given in a split dose (30/mg/kg each) separated by 3 hours. The agent was gel encapsulated to reduce appreciation of odor and taste and mimic appearance of the placebo.
Period: Overall Study
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Started | 184 | 186
Completed | 183 | 183
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo Control at 12-16 Weeks Gestation: Placebo was made with the same color-coded gelatin capsules with the inert compound dextrose.
- Praziquantel at 12-16 Weeks Gestation: Praziquantel was administered orally as 60 mg/kg given in a split dose (30/mg/kg each) separated by 3 hours.
- Total: Total of all reporting groups
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation | Total
Number analyzed (Participants) | 184 | 186 | 370
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 186 | 370
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.3) | 26.2 (6.6) | 26.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 186 | 370
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Philippines | 184 | 186 | 370

OUTCOME MEASURES:

1. Primary Outcome: Mean Newborn Birth Weight
Description: Birth weight was collected for live infants at the time of delivery by a trained midwife, or within 24 hours of delivery for participants who chose to deliver at home with a helot, a birth attendant without formal training.
Time Frame: Within 24 hours of delivery.
Population: All newborns for whom birth weights were reported were included in the analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 181 | 180
kilograms | 2.85 (0.39) | 2.85 (0.44)
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.988, t-test, 2 sided — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

2. Secondary Outcome: Number of Participants Whose Pregnancy Resulted in a Live Birth
Description: Each participant was followed until delivery to record if the outcome of the pregnancy was a live birth. Live births were defined as the complete expulsion or extraction from its mother of a product of conception, irrespective of the duration of the pregnancy, which, after such separation, breathes or shows any other evidence of life such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles, whether the umbilical cord had been cut or the placenta was attached.
Time Frame: At delivery
Population: All participants for whom the status of the infant at delivery was reported are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 183
participants | 181 | 181
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p > 0.999, Chi-squared — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

3. Secondary Outcome: Mean Change in Maternal Hemoglobin From 14 to 32 Weeks Gestation
Description: Hemoglobin concentration in a venous blood sample collected at 14 and 32 weeks gestation was measured using a multi-analyte analyzer. Each participant's change in hemoglobin concentration between the two timepoints was determined, and the mean and standard deviation for each group calculated.
Time Frame: 14 weeks and 32 weeks gestation
Population: All participants for whom hemoglobin concentrations were reported are included in the analysis.
Measure: Mean (Standard Deviation); unit: grams/deciliter
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
grams/deciliter | -0.42 (1.39) | -0.44 (1.38)
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.926, t-test, 2 sided — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

4. Secondary Outcome: Median Change in Maternal Transferrin Receptor:Ferritin Ratio From 14 to 32 Weeks Gestation
Description: To assess total body iron, one needs to assess the storage compartment, which will contain sequestered iron, and the functional compartment, which represents bioavailable iron. Body iron status is defined by the two laboratory measurements that reflect these compartments, ferritin and serum transferrin receptor. The serum transferrin receptor:ferritin ratio has been shown in quantitative phlebotomy studies to provide an accurate assessment of total body iron over the entire range of status. At 14 and 32 weeks gestation, a blood sample was collected for assessment of total body iron by determination of the transferrin receptor:ferritin ratio. Each participant's change in ratio was calculated, and the median and interquartile range were determined for each group.
Time Frame: 14 weeks and 32 weeks gestation
Population: All participants for whom transferrin receptor:ferritin ratio was reported at both timepoints are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
ratio | 0.0 (75.88) [0.0 to 15.47] | 0.0 (162.4) [0.0 to 7.56]
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.502, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

5. Secondary Outcome: Median Maternal Hepcidin at 32 Weeks Gestation
Description: Anemia of inflammation was assessed via maternal urine hepcidin levels. In response to inflammation, elevated serum levels of hepcidin is synthesized. Hepcidin causes sequestration of iron from bio-available forms to storage forms such as ferritin and decreases intestinal absorption of iron. Hepcidin was measured in participants' urine at 32 weeks gestation.
Time Frame: 32 weeks gestation
Population: All participants for whom hepcidin levels were reported are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: nanograms/milliliter
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
nanograms/milliliter | 2.58 (5.06) [0.94 to 6.00] | 3.38 (4.32) [1.18 to 5.50]
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.439, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

6. Secondary Outcome: Mean Change in Maternal Weight From 14 to 32 Weeks Gestation
Description: Maternal weight gain was assessed by measuring participants' weight in kilograms. The weight increase from 14 to 32 weeks was determined for each participant, and the mean and standard deviation calculated.
Time Frame: 14 and 32 weeks gestation
Population: All participants for whom weight was reported at both timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
kilograms | 0.33 (0.13) | 0.32 (0.13)
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.704, t-test, 2 sided — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

7. Secondary Outcome: Mean Change in Maternal Thigh Skinfold Thickness From 14 to 32 Weeks Gestation
Description: Maternal fat stores were measured by thigh skinfold thickness obtained using a Holtain skinfold caliper. The thickness increase from 14 to 32 weeks was determined for each participant, and the mean and standard deviation calculated.
Time Frame: 14 and 32 weeks gestation
Population: All participants for whom thigh skinfold thickness was reported at both timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
millimeters | 0.08 (0.09) | 0.08 (0.09)
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.517, t-test, 2 sided — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

8. Secondary Outcome: Newborn Median Serum Transferrin Receptor:Ferritin Ratio
Description: To assess total body iron, the serum transferrin receptor:ferritin ratio was assessed in the infant. At delivery, a heel stick blood sample and a cord blood sample were collected for assessment of total body iron by determination of the transferrin receptor:ferritin ratio.
Time Frame: 0-6 days after delivery.
Population: All infants for whom transferrin receptor and ferritin were reported are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 181 | 181
ratio
  Cord Blood | 1.76 (480.39) [0.00 to 5.29] | 1.33 (1392.55) [0.00 to 4.36]
  Heel Stick | 0.00 (239.81) [0.00 to 0.10] | 0.00 (162.24) [0.00 to 0.00]
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Analysis included the transferrin receptor: ferritin ratio from the cord blood; Test type: Superiority or Other; p = 0.524, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05
Statistical Analysis 2: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Analysis included the transferrin receptor: ferritin ratio from the heel stick; Test type: Superiority or Other; p = 0.070, Wilcoxon (Mann-Whitney) — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

9. Secondary Outcome: Number of Subjects With Reduction in S. Japonicum Egg Counts From Screening to 22 Weeks Gestation of Greater Than 90 Percent
Description: Parasitologic response to treatment was evaluated by counting S. japonicum eggs per gram of stool at screening and again at 22 weeks gestation. Success of treatment was pre-specified as greater than 90 percent reduction in egg count from screening to 22 weeks gestation.
Time Frame: Screening and 22 weeks gestation
Population: All participants for whom egg counts were reported are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 184 | 184
participants | 92 | 157
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p < 0.001, Chi-squared — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

10. Secondary Outcome: Number of Participants Reporting Serious Adverse Events Within 24 Hours of Dosing
Description: Participants were observed in hospital for 24 hours after dosing for serious adverse events. Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof (for reasons other than the 24-hour observation period); resulted in a congenital anomaly/birth defect; or may have jeopardized the participant, or required intervention to prevent one of these outcomes.
Time Frame: Within 24 hours of dosing
Population: All participants were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 184 | 186
participants | 0 | 0

11. Secondary Outcome: Number of Participants Experiencing Fetal Loss by Abortion
Description: Abortion was defined by the protocol as bleeding followed by fetal loss as supported by ultrasound before 20 weeks gestation. Abortion was an important safety outcome measure due to the fact that abortion would occur closer to the time of dosing than miscarriage or stillbirth. Participants were observed in hospital for 24 hours after dosing and asked to return for any bleeding at any time.
Time Frame: After dosing and before 20 weeks gestation
Population: All participants were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 184 | 186
participants | 0 | 0

12. Secondary Outcome: Number of Participants Reporting Abnormalities in Hematology Assessments Within 24 Hours of Dosing
Description: Toxicity to maternal bone marrow, kidney, and liver was assessed by laboratory parameters collected just before and 24 hours after dosing. Specifically, blood was drawn just before the dose at 12-16 weeks gestation to determine baseline complete blood count, including white blood count (WBC), platelets, and hemoglobin. Blood was then drawn 24 hours after the second part of the split dose and before discharge from the hospital to assess any changes in these parameters. White blood count was abnormal at or above 10,800 or at or below 3500 cells/square millimeter (sq mm), platelets were abnormal at or below 140,000 cells/sq mm, and hemoglobin was abnormal at or below 10.9 grams/deciliter (g/dL).
Time Frame: Just before and 24 hours after dosing
Population: All participants were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 184 | 186
participants
  White Blood Cell Abnormal | 69 | 60
  Platelets Abnormal | 3 | 0
  Hemoglobin Abnormal | 54 | 56

13. Secondary Outcome: Number of Participants Reporting Abnormalities in Clinical Chemistry Assessments Within 24 Hours of Dosing
Description: Toxicity to maternal kidney and liver was assessed by laboratory parameters collected just before and 24 hours after dosing. Specifically, blood was drawn just before the dose at 12-16 weeks gestation to determine baseline blood urea nitrogen (BUN), creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and bilirubin. Blood was then drawn 24 hours after the second part of the split dose and before discharge from the hospital to assess any changes in these parameters. Any values that were 1.1 times the upper limit of normal or greater for the parameter were considered abnormal.
Time Frame: Just before and 24 hours after dosing
Population: All participants were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 184 | 186
participants
  Blood Urea Nitrogen (BUN) Abnormal | 127 | 137
  Creatinine Abnormal | 23 | 39
  Aspartate Aminotransferase (AST) Abnormal | 8 | 9
  Alanine Aminotransferase (ALT) Abnormal | 13 | 10
  Bilirubin Abnormal | 127 | 137

14. Secondary Outcome: Number of Participants Whose Infant Was Born With Congenital Anomalies
Description: The newborn was examined by the midwife at delivery and within 2-6 days of delivery to assess the presence of congenital anomalies and well-being. The newborn was also examined by study pediatrician at 28 days of life.
Time Frame: At delivery, within 2-6 days of delivery, and at 28 days
Population: All newborns are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 181 | 181
participants | 1 | 1
Statistical Analysis 1: Comparison: Placebo Control at 12-16 Weeks Gestation vs Praziquantel at 12-16 Weeks Gestation; Test type: Superiority or Other; p = 0.991, Chi-squared — The p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

15. Secondary Outcome: Number of Participants With Pre-eclampsia
Description: Participants were assessed for the presence of pre-eclampsia at both the 22 and 32 week visits. Pre-eclampsia was defined by the presence of proteinurea (2+ protein on urine dipstick) and a single diastolic blood pressure reading of 100 millimiters of mercury (mm Hg) or above OR more than one reading, four hours apart, of 90 mm Hg or above.
Time Frame: 22 weeks and 32 weeks
Population: All participants seen at both timepoints are included.
Measure: Number; unit: participants
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 183 | 181
participants | 0 | 0

16. Secondary Outcome: Maternal Serum Cytokine Levels of TNF-alpha, TNF-alpha Receptors I and II, IL-1, and IL-6
Description: Extra-placental mechanisms mediating improved outcomes in the PZQ group were planned to be evaluated with maternal serum cytokine levels, particularly TNF-alpha, TNF-alpha receptors I and II, IL-1, and IL-6. These assays were intended to be performed only if the primary objective of the study was met; therefore, there will be no results reported for this outcome measure.
Time Frame: At 32 weeks gestation
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Placental Blood Cytokine Levels
Description: Cytokine assays were planned to be performed with culture supernatant harvested from placental explant cultures. The cytokines were to be measured with a multi-analyte analyzer. These assays were intended to be performed only if the primary objective of the study was met; therefore, there will be no results reported for this outcome measure.
Time Frame: At delivery
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Cytokeratin 18 Neo-epitope Staining as a Measure of Apoptosis
Description: A study hypothesis was that peripheral serum obtained from S. japonicum infected, treated mothers would induce a lower level of apoptosis (programmed cell death) in cultured trophoblasts as measured by cytokeratin 18 neo-epitope staining compared to peripheral serum obtained from S. japonicum infected, PZQ untreated mothers. This assay was planned to be completed only if the primary objective was met; therefore, there will be no data for this outcome measure.
Time Frame: 32 weeks gestation
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Praziquantel Pharmacokinetic Concentrations
Description: Two plasma samples were collected during the overnight hospitalization from approximately 200 subjects that remained at the time of study modification to incorporate PK studies. Subjects had samples collected based on one of two sample collection strategies: 4.5 and 8 hr after the first praziquantel dose or 6 and 10 hr after the first praziquantel dose. Subjects randomized to an even study number were assigned to the 4.5 and 8 hour schedule. Subjects randomized to an odd study number were assigned to the 6 and 10 hour schedule. Samples only from subjects randomized to receive praziquantel were analyzed for praziquantel. Samples drawn from subjects randomized to the control group were not analyzed. Praziquantel concentrations (ng/ml) were assayed using high performance liquid chromatography-electrospray mass spectrometry in the University of California at San Diego Pediatric Clinical Pharmacology Laboratory.
Time Frame: 4.5 and 8 hours after the first praziquantel dose (subjects assigned to an even study number) or 6 and 10 hours after the first praziquantel dose (subjects assigned to an odd study number).
Population: The analysis population for pharmacokinetics descriptive analyses was defined as all subjects who had plasma samples collected and who were randomized to receive PZQ (N=99; 50 subjects at 4.5 and 8 hr after first PZQ dose and 49 at 6 and 10 hr after first PZQ dose).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 99
ng/mL
  4.5 Hours, n=50 | 814.7 [289.8 to 1580.6]
  6 Hours, n=49 | 945.2 [362.0 to 1365.0]
  8 Hours, n=50 | 687.8 [107.7 to 1137.6]
  10 Hours, n=49 | 422.2 [50.5 to 769.1]

20. Secondary Outcome: 4-hydroxy Praziquantel Pharmacokinetic Concentrations
Description: Since pregnancy is associated with increased cytochrome P450 activity and physiologic changes in the gastrointestinal tract that tend to reduce drug absorption, praziquantel pharmacokinetics may be affected by pregnancy. Thus, the metabolite-to-parent drug ratio may serve as a differential marker to help determine if variability in drug exposure following oral administration during pregnancy is due to altered metabolism or drug absorption. Samples that were collected from subjects who were randomized to receive praziquantel were analyzed for praziquantel and 4-hydroxy praziquantel concentrations. Assays were performed using high performance liquid chromatography-electrospray mass spectrometry in the University of California at San Diego Pediatric Clinical Pharmacology Laboratory. Descriptive statistics were obtained for concentrations at each of the four sparse sampling timepoints.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Praziquantel at 12-16 Weeks Gestation
Number analyzed (Participants) | 99
ng/ml
  4.5 Hours, n=50 | 4020.1 [2022.1 to 5846.6]
  6 Hours, n=49 | 4590.8 [2982.5 to 7514.5]
  8 Hours, n=50 | 5373.7 [1476.6 to 7503.2]
  10 Hours, n=49 | 4304.1 [994.2 to 6344.3]

ADVERSE EVENTS:
Time Frame: Solicited systemic symptoms were observed in clinic 24 hours after treatment and recorded for 14 days post treatment. Unsolicited adverse events and SAEs were evaluated at clinic visits and passively reported through 28 days post delivery.
Description: For solicited symptoms recorded on the Memory Aid in the 14 days after treatment, a participant was considered to have one event if it was reported as experienced at any time in the 14-day period.
Arm/Group | Placebo Control at 12-16 Weeks Gestation | Praziquantel at 12-16 Weeks Gestation
Serious Adverse Events (participants affected / at risk) | 34/184 | 45/186
Other Adverse Events (participants affected / at risk) | 159/184 | 176/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Control at 12-16 Weeks Gestation (N=184) | Praziquantel at 12-16 Weeks Gestation (N=186)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Amoebiasis (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 5 (6) | 4 (4)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
17-hydroxyprogesterone increased (Investigations) | 1 (1) | 0 (0) — Reported in infant born to participant
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) — Reported in infant born to participant
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) — Reported in infant born to participant
Chemical injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Reported in infant born to participant
Cleft lip and palate (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) — Reported in infant born to participant
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1) — Reported in infant born to participant
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — Reported in infant born to participant
Glucose-6-phosphate dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 4 (4) — Reported in infant born to participant
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) — Reported in infant born to participant
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 1 (1) — Reported in infant born to participant
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Reported in infant born to participant
Jaundice (Hepatobiliary disorders) | 2 (2) | 1 (1) — Reported in infant born to participant
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Reported in infant born to participant
Microtia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) — Reported in infant born to participant
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Reported in infant born to participant
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Reported in infant born to participant
Neonatal pneumonia (Infections and infestations) | 2 (2) | 5 (5) — Reported in infant born to participant
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Reported in infant born to participant
Omphalitis (Infections and infestations) | 1 (1) | 0 (0) — Reported in infant born to participant
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) — Reported in infant born to participant
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Reported in infant born to participant
Premature baby (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2) — Reported in infant born to participant
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Reported in infant born to participant
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) — Reported in infant born to participant
Talipes (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) — Reported in infant born to participant
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — Reported in infant born to participant
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Control at 12-16 Weeks Gestation (N=184) | Praziquantel at 12-16 Weeks Gestation (N=186)
Anaemia (Blood and lymphatic system disorders) | 51 (52) | 47 (48)
Abdominal pain lower (Gastrointestinal disorders) | 15 (16) | 12 (12)
Pyrexia (General disorders) | 13 (14) | 16 (17)
Nasopharyngitis (Infections and infestations) | 7 (8) | 15 (16)
Urinary tract infection (Infections and infestations) | 13 (13) | 10 (11)
Blood pressure increased (Investigations) | 10 (10) | 3 (3)
Haemoglobin decreased (Investigations) | 16 (17) | 9 (9)
Urine leukocyte esterase positive (Investigations) | 10 (10) | 4 (4)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 15 (16) | 10 (10)
Dysuria (Renal and urinary disorders) | 4 (4) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (41) | 37 (40)
Pyrexia (General disorders) | 47 (47) | 39 (39) — This symptom was solicited as the oral temperature taken by the subject daily for 14 days. Oral temperatures were graded during statistical analyses to define pyrexia as an oral temperature of 37.5 degrees Celsius or greater on any of the 14 days.
Headache (Nervous system disorders) | 82 (82) | 99 (99)
Malaise (General disorders) | 68 (68) | 81 (81)
Abdominal Pain (Gastrointestinal disorders) | 63 (63) | 76 (76)
Nausea (Gastrointestinal disorders) | 68 (68) | 94 (94)
Vomiting (Gastrointestinal disorders) | 53 (53) | 77 (77)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 14 (14) — Dyspnoea was solicited as 'shortness of breath'.
Dizziness (Nervous system disorders) | 50 (50) | 100 (100)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less